CLINICAL TRIAL: NCT00697073
Title: A Phase III Open-Label, Single Group Extension Study of the Safety and Tolerability of Idebenone in the Treatment of Friedreich's Ataxia Patients
Brief Title: Study to Assess the Safety and Tolerability of Idebenone in the Treatment of Friedreich's Ataxia Patients
Acronym: IONIA-E
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNT-III-002-E
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Results first posted 2011-08-04 (Estimated); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Friedreich's Ataxia
Keywords: Friedreich's Ataxia; Idebenone; ICARS
MeSH Terms: conditions — Friedreich Ataxia | interventions — idebenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): high dose Idebenone
  Interventions: Drug: Idebenone

INTERVENTIONS:
Drug: Idebenone — Patients ≤ 45 kg/99 lbs: idebenone 1350 mg/day; Patients > 45 kg/99 lbs: idebenone 2250 mg/day

SUMMARY:
This study is meant to assess the safety and tolerability of idebenone in patients with Friedreich's Ataxia over a 12 months period.

DETAILED DESCRIPTION:
The study involves 6 clinic visits.

ELIGIBILITY:
Inclusion criteria:

* Friedreich's ataxia patients completing core study SNT-III-002 (NCT00537680) and presenting at Week 24 (Visit 5) of that study
* Body weight ≥ 25kg/55 lbs
* Negative urine pregnancy test
* Patients who in the opinion of the investigator are able to comply with the requirements of this study

Exclusion criteria:

* Adverse events during the course of SNT-III-002(NCT00537680)which in the opinion of the investigator are attributable to idebenone and preclude further treatment with idebenone
* Clinically significant abnormalities of clinical hematology or biochemistry including, but not limited to, elevations greater than 2 times the upper limit of normal of AST, ALT or creatinine
* Treatment with coenzyme Q10, vitamin E (if taken at a dose 5 times above the daily requirement) or other sources of idebenone within the past month
* Parallel participation in another clinical drug trial
* Past or present history of abuse of drugs or alcohol
* Pregnancy or breast-feeding

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Perlman, MD, Principal Investigator — University of California, Los Angeles; David Lynch, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - David Geffen School of Medicine, UCLA, Los Angeles, California
  - The Children's Hopsital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Meier T, Perlman SL, Rummey C, Coppard NJ, Lynch DR. Assessment of neurological efficacy of idebenone in pediatric patients with Friedreich's ataxia: data from a 6-month controlled study followed by a 12-month open-label extension study. J Neurol. 2012 Feb;259(2):284-91. doi: 10.1007/s00415-011-6174-y. Epub 2011 Jul 22. PMID 21779958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 59 subjects completed the study. Nine subjects did not complete the study. However, neurological efficacy data (ICARS, FARS) are available for Week 52 from 61 patients.
  All 68 subjects enrolled in this study were included in the Safety population.
Groups:
- High Dose Idebenone: Patients ≤ 45 kg/99 lbs: idebenone 1350 mg/day (3 x 150 mg tablets, t.i.d.)
  Patients > 45 kg/99 lbs: idebenone 2250 mg/day (5 x 150 mg tablets, t.i.d.)
Period: Overall Study
Arm/Group | High Dose Idebenone
Started | 68
Completed | 59
Not Completed | 9
Not completed — Withdrawal by Subject | 2
Not completed — Pregnancy | 1
Not completed — non compliance and other | 6

BASELINE CHARACTERISTICS:
Arm/Group | High Dose Idebenone
Number analyzed (Participants) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 68
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.0 (2.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 68

OUTCOME MEASURES:

1. Primary Outcome: Change in ICARS
Description: International Cooperative Ataxia Rating Scale (ICARS):
  ICARS consists of a one-hundred-point semi-quantitative scale based upon 19 simple testing manoeuvres compartmentalized into postural and stance disorders, limb ataxia, dysarthria and oculomotor disorders and has been previously used in this patient population with good inter-rater reliability.
  A total score of 0 points represents the best possible score, and a value of 100 points is the worst possible score. Therefore, a negative change in ICARS score represents an improvement. A higher score also indicates more disability.
Time Frame: baseline and 12 months
Population: A total of 59 subjects completed the study. Nine subjects did not complete the study. However, neurological efficacy data (ICARS, FARS) are available for Week 52 from 61 patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Dose Idebenone
Number analyzed (Participants) | 61
units on a scale | 1.1 (5.64)

2. Secondary Outcome: FARS (Friedreich's Ataxia Rating Scale)
Description: FARS consists of a 25 manoeuvre exam along with 4 quantitative performance measures. The neurological exam covers bulbar function, upper limb coordination, lower limb coordination, peripheral nervous system function, deep tendon reflexes, stability and gait. The use of FARS has been recently validated as a sensitive scale for this population. The FARS consists of three subscales, comprising a general score for ataxia, a score for activities of daily living (ADL) and a neurological examination. The scores can be added to make a total score ranging from 0 to 159. A higher score indicates a greater level of disability.
Time Frame: baseline and 12 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Dose Idebenone
Number analyzed (Participants) | 61
units on a scale | 2.3 (5.59)

3. Secondary Outcome: Nature of Adverse Events
Time Frame: 12 Months
Population: All 68 subjects enrolled in this study were included in the Safety population.
Measure: Number; unit: events
Arm/Group | High Dose Idebenone
Number analyzed (Participants) | 68
events
  Infections and Infestations | 117
  Gastrointestinal Disorders | 97
  Musculoskeletal and Connective Tissue Disorders | 75

4. Secondary Outcome: Frequency/Number of Mild, Moderate, and Severe Adverse Events
Time Frame: 12 months
Population: All 68 subjects enrolled in this study were included in the Safety population.
Measure: Number; unit: events
Arm/Group | High Dose Idebenone
Number analyzed (Participants) | 68
events
  mild | 30
  moderate | 32
  severe | 4

ADVERSE EVENTS:
Arm/Group | High Dose Idebenone
Serious Adverse Events (participants affected / at risk) | 4/68
Other Adverse Events (participants affected / at risk) | 66/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Idebenone (N=68)
cardiac failure (Cardiac disorders) | 1 (1)
tachycardia (Cardiac disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypotension (General disorders) | 1 (1)
Deep vein thrombosis (General disorders) | 1 (1)
Dehydratation (General disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
intra uterine death (Pregnancy, puerperium and perinatal conditions) | 1 (1)
abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Idebenone (N=68)
headache (General disorders) | 21
upper respiratory tract infection (Infections and infestations) | 18
nausea (Gastrointestinal disorders) | 15
pyrexia (General disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No